CLINICAL TRIAL: NCT06482216
Title: Correlation of Protection Against Varicella in an Exploratory Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-VZV-4007
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vaccination group: The last dose of varicella vaccine given 30 days before enrollment was manufacture by Sinovac (Dalian) Vaccine Technology Co. LTD.,(Sinovac).
  Interventions: Biological: Varicella vaccine
- Non-vaccination group: Without varicella vaccine history

INTERVENTIONS:
Biological: Varicella vaccine — lyophilized powder,subcutaneous injection
  Groups: Vaccination group

SUMMARY:
This study consists of two parts. Part 1 is a retrospective cohort study and part 2 is a prospective cohort study. In Part 1 ,the scaled logit model was used to assess the correlation between varicella-zoster virus (VZV) antibody titers using fluorescent-antibody-to-membrane-antigen assay (FAMA) 30 days after varicella vaccine immunization and the risk of subsequent varicella breakout/disease , to determine the protective threshold for achieving FAMA antibodies. Part 2 was to validate the model in part 1.

DETAILED DESCRIPTION:
Part 1 was based on a previous Phase Ⅲ, randomized, placebo-controlled clinical trial (NCT02981836) conducted from 2016 to 2017. The analysis data of part 1 was from historical serum, historical varicella cases and additional one year case monitoring conducted as an extension of the Phase III study.

Part 2 was conducted based on close contacts of varicella cases. All close contacts without varicella symptoms will be recruited and followed up for 14 days to monitor the occurrence of the varicella cases. Part 2 aimed to compare the differences of FAMA antibody titers in varicella breakthrough cases, non-breakthrough cases, and non-cases at the time of exposure to validate/calibrate the model established in part 1.

ELIGIBILITY:
Inclusion Criteria:

* 1-12 years children who were the siblings or children of the indicator varicella cases, or the deskmates/roommates of the indicator varicella cases;
* Having close contacts with the indicator varicella cases at least 2 days during the period from 5 days before the onset and 2 days after the onset;
* Without varicella vaccination history or having varicella vaccination history (the last dose of varicella was manufacured by Sinovac, with an interval of >30 days before enrollment)
* Subjects/legal guardian can understand and sign the informed consent;
* Being able to provide legal proof of identity.

Exclusion Criteria:

* Without varicella history;
* Body temperature ≥37.0℃ on the day of enrollment, or skin rash on the head, torso, and limbs;
* Having any confirmed or suspected immunodeficiency disorder, including tumor patients undergoing chemotherapy, human immunodeficiency virus (HIV) infection, continuous use of steroid hormones for more than 30 days (prednisone equivalent ≥2mg/kg days in children), or having other immunosuppressive disorder as determined by the clinician;
* The investigators considered that participation in this study was not appropriate for various other reasons.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: There was no inclusion/exclusion criteria in the retrospective cohort study. The inclusion/exclusion criteria were only applicable in the prospective cohort.
  Subjects in the retrospective cohort study aged 8-20 years were from a previous phase Ⅲ study. There is no limit to the sample size of the retrospective cohort, which is based on the number of final follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2027-05-10 (Estimated); Study Completion 2028-10-10 (Estimated)

PRIMARY OUTCOMES:
Retrospective cohort: Varicella confirmed case | one year after enrollment
  Varicella confirmed case during an additional year follow-up period (pooled with varicella confirmed case from previous phase Ⅲ study)
Retrospective cohort: Varicella antibody titer | on Day 30 after vaccination
  Varicella antibody titer on Day 30 after vaccination (historical serum)
Prospective cohort: Varicella confirmed case | Within 14 days after enrollment
  Varicella confirmed case during the 14-day follow-up period
Prospective cohort: Varicella antibody titer | Enrollment
  Varicella antibody titer on exposure

SECONDARY OUTCOMES:
Prospective cohort: Varicella antibody titer | Within 3 days after eruption
  Varicella antibody titer in the acute period of varicella confirmed case
Prospective cohort: Varicella antibody titer | Within 14-21 days after eruption
  Varicella antibody titer in the convalescent period of varicella confirmed case

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Liu, Principal Investigator — Yunnan Provincial Center for Disease Control and Prevention; Zhiqiang Xie, Principal Investigator — Henan Provincial Center for Disease Control and Prevention

IPD SHARING:
Plan to Share IPD: No